CLINICAL TRIAL: NCT00268827
Title: A Comparison of Adverse Events and Quality of Life Before and After Switching From Kaletra Soft-Gel Capsules (SGC) to Kaletra Tablets in an African American Cohort
Brief Title: A Comparison Study of Kaletra Soft-Gel Capsules and Kaletra Tablets in an African American Cohort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AIDS Arms Inc. (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 70-1002-070; 371-11-05
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: HIV-1; AIDS
Keywords: Kaletra; Comparison; Quality of Life; African American
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Kaletra soft-gel capsules switched to Kaletra tablets
Device: MOS-HIV Health and Medication Satisfaction Survey, Global Conditioning Improvement and Therapy Preference Questionnaire

SUMMARY:
The purpose of this study is to compare Kaletra tablets with Kaletra soft-gel capsules to see if there is any change in the side effects you may have and to see how people in the study feel about using the tablets.

DETAILED DESCRIPTION:
The demand for once-a-day easily tolerated therapies is increasing. While Abbott Laboratories 418 study has demonstrated the efficacy of Kaletra® with both BID and QD dosing with capsules, the pill count of QD dosing may decrease its attractiveness for this population. In some patients, issues such as diarrhea, nausea, food restrictions, or the need to refrigerate their medication may also impact quality of life and possibly lead to non adherence and ultimately treatment failure. Moreover, it is believed that the diarrhea associated with Kaletra® capsules may be the result of capsule excipients that are unrelated to the active drug.

Kaletra® has a long track record of being highly potent and not selective for protease inhibitor resistance as evidence by the Phase II Study 720. The results of this study demonstrate that ABT-378/ritonavir therapy is highly potent, durable, and well tolerated when administered concomitantly with two nucleoside analog reverse transcriptase inhibitors to antiretroviral-naïve HIV-1 infected individuals. A high proportion of subjects achieved normal viral suppression (< 50 copies/ml - 78% by ITT). No discontinuations due to study drug -related clinical or laboratory adverse events occurred during the first 48 weeks of study but the most common adverse effect was diarrhea (25%). Given the high oleic content of the capsules, dosing all six capsules at once may cause a "bolus" of this acid leading to increased diarrhea. Because of the viral suppression advantages, there is desire to see if there is a difference in quality of life and tolerability between the soft-gel capsules and the new tablet formulation of Kaletra® which allows for fewer tablets per day and does not include additives possibly associated with increased diarrhea.

Study MOO-267 (PLATO), a multi-center study evaluated and demonstrated improved quality of life when switching from other regimens (efavirenz, nevirapine, indinavir, and nelfinavir) to Kaletra®. Instruments used to measure change in quality of life included the AIDS Clinical Trial Group (ACTG) Symptom Distress Module (ASDM) which measures the presence of bothersome symptoms commonly seen with HIV and ARV treatment; the Medical Outcomes Study-HIV Health Survey (MOS-HIV) which is widely used to evaluate the Quality of Life (QOL) of HIV infected patients; and the Center for Epidemiological Studies and Depression (CES-D), a validated self-reporting questionnaire used as a screening tool for depression.

The hypothesis is that patient's quality of life will improve when switched from Kaletra® soft-gel to Kaletra® tablets. The tablet formulation of Kaletra® will improve quality of life by simplifying current HAART regimens by decreasing pill count, improving tolerability, eliminating food restrictions and the need for drug refrigeration. African-American subjects were selected for this study because they are an understudied population and due to adherence behavior. In reviewing Abbott Study 418 and Study MOO 267 the percent of African-American enrollees accounted for 27% and 15% of the study groups respectively.1,4 In studies where there is an association between socio demographic factors and adherence behavior, the direction is consistent: younger age, non-white race, lower income, lower literacy and unstable housing was associated with non-adherence. Adherence behavior refers to the extent to which patients take their medication as prescribed by their health provider. As stated above, patients who are younger, non white race, lower income and live in unstable housing are less likely to adhere to the prescribed medication regime. It is important to evaluate antiretroviral therapy formulations to validate patient tolerability and acceptance in order to promote drug adherence. This study will compare the tolerability and acceptance of patients on Kaletra® soft-gel capsules with that of Kaletra® tablet formulation utilizing validated instruments as described above.

ELIGIBILITY:
Inclusion Criteria:1. African American male or female patients ≥ 18 years of age 2. Documented HIV-infected 3. Currently on Kaletra® soft-gel capsules for >2 weeks 4. Competent and willingness to sign and date a written informed consent 5. No recent acute illness in the preceding 30 days which in the opinion of the investigator would preclude inclusion in the study 6. No current gastrointestinal symptoms at baseline of grade II or greater 7. A female is eligible to enter and participate in this study if she is of:

* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal) or
* Child-bearing potential, has a negative urine or serum pregnancy test at screen, and agrees to one of the following:
* Complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and for at least 2 weeks after completion or premature discontinuation from the study to account for elimination of the investigational drug. Should a patient decide to become sexually active during the course of the study, she must be counseled and be willing to use one of the birth control methods listed below:
* Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide)
* Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion)
* Sterilization (female patient or male partner of female patient)
* Any other methods with published data showing that the lowest expected failure rate for that method is <1% per year.

NOTE: Data are insufficient to exclude a clinically important interaction of LPV/r with drugs, such as hormonal contraceptives, that are highly metabolized by the cytochrome P450 enzyme system. As a result, hormonal contraception is not considered adequate.

Exclusion Criteria:1. Positive pregnancy test or breast-feeding 2. Known hypersensitivity to study medications 3. Inability to conform to protocol procedures, including alcohol or drug abuse, untreated psychiatric illness 4. An unwillingness or presence of any condition that will impair the ability to swallow medications 5. Patient has required treatment with radiation therapy or cytotoxic chemotherapeutic agents within 4 weeks prior to entry, or has an anticipated need for these agents within the study period.

6. Patient requires treatment with immunomodulating agents, such as systemic corticosteroids, interleukins, or interferon's within 4 weeks prior to study entry, or patients who have received an HIV immunotherapeutic vaccine within 3 months prior to entry.

7. Patient requires inhaled or intranasal fluticasone

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-12; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To compare the tolerability and acceptance of patients on the Kaletra® soft gel with that of Kaletra® tablet formulation utilizing the Symptoms Distress Module developed by the ACTG and the Center Epidemiological S

SECONDARY OUTCOMES:
Proportion of subjects maintaining or achieving HIV-RNA < 400 or < 50 copies/ml, maintaining or increasing CD4 T-lymphocyte count;G.I. or other adverse events grade 2-4;Other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Marsden K. Rawlings, MD, Principal Investigator — AIDS Arms Inc./Peabody Health Center
Locations (1):
- AIDS Arms Inc./Peabody Health Center, Dallas, Texas, United States